CLINICAL TRIAL: NCT05931159
Title: Effects of Abdominal Hypopressive Exercises on Diastasis Recti in Postpartum Women
Brief Title: Effects of AHEs on DrA in Postpartum Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01538 Fatima Iftikhar
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Diastasis Recti
Keywords: Diastasis Recti; Diastasis Recti and weakness of Linea alba; Low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominal Hypopressive Training (Experimental): The Abdominal hypopressive Exercises along with home plan based on conventional exercises.
  Interventions: Other: Abdominal Hypopressive Training
- Conventional Physical therapy for DrA (Active Comparator): Draw-in maneuver in supine, quarduped, prone lying, bent leg fall outs, curl ups, and front and side planks.
  Interventions: Other: Conventional Physical therapy for DrA

INTERVENTIONS:
Other: Abdominal Hypopressive Training — Week 1 and 2 - Patient education , Hypopressive Maneuvers in Standing, Sitting and Supine 5-7 repetitions x 5 sets, with a 10-second hold each time, rest for 30 seconds between each set, 2 days/week.
  Week 3 and 4, Hypopressive breathing in with varying arm movements along with Week 1 and 2 protocols.
  Week 5 to 8 - Hypopressive breathing in kneeling, Four-point kneeling and sitting, and supine positions with varying arm movements 5-7 repetitions x 5 sets, with a 10-second hold each time, rest for 30 seconds between each set, 2 days/week.
  Arms: Abdominal Hypopressive Training
Other: Conventional Physical therapy for DrA — Week 1 to 4, Draw-in maneuver in supine, Quadruped and Prone lying, Bent knee Fallouts and Curl ups. (8 to 12 repetitions x 3 sets, 2 days/week)
  Week 5 to 8, Front and side planks added to week 1 to 4 exercises. (12 to 20 repetitions x e sets, 2 days/week)
  Arms: Conventional Physical therapy for DrA

SUMMARY:
This study is aimed to determine the effects of Abdominal Hypopressive exercises on IRD, Lumbopelvic pain, Body Image and abdominal muscle function in postpartum women.

DETAILED DESCRIPTION:
Postnatal women wish to resume abdominal exercises shortly after delivery to improve trunk function and restore the pre-pregnant state of the body. Diastasis recti is a common occurrence in the postpartum period which is associated with both physical impairments and body image concerns. Despite the high prevalence, treatment options are still being explored to identify the best approach to resolve it. Exercise is a conservative method to reduce IRD and improve the associated symptoms and quality of life of postpartum females. Most of the previous studies have used either digital nylon calipers or digital palpation methods for the outcome assessment of DrA which has important implications. Fewer studies have used the gold standard US diagnosis. Despite various studies being conducted on the effect of exercise on DrA, the results are still nonconclusive with a deficiency of a standardized protocol. Multifaceted and clinically meaningful assessments have been proposed to be investigated by the previous literature.

ELIGIBILITY:
Inclusion Criteria:

* 12 weeks to 36 weeks postpartum
* Both vaginal delivery and C-section
* Lumbopelvic pain (NPRS >4)
* Diagnosis of DrA by calliper: 3 cm below the umbilicus: >22 mm, at the umbilicus: >20 mm, 3 cm above the umbilicus: >14 mm
* Primiparous females

Exclusion Criteria:

* Any conditions affecting the ability to perform exercise or activity of daily living.
* Previous spinal or abdominal surgery, and neuromuscular diseases.
* Severe DrA >5cm with the herniation or requiring surgical repair.
* LBP associated with disc herniation, spondylolysis, and degenerative changes of the spine

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 38 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Inter Recti Distance | 8th Week
  Changes from baseline Ultrasound imaging (US) is the gold standard for IRD assessment. USI is an accurate and valid method of measuring IRD size and location. Patient will be graded as having an IRD of > 22 mm, 3 cm below the umbilicus OR > 20 mm at the umbilicus OR >14 mm, 3 cm above the umbilicus.
Lumbopelvic Pain | 8th Week
  Changes from baseline The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. Zero usually represents 'no pain at all' whereas the upper limit of 10 represents 'the worst pain ever possible'.
The Oswestry Disability Index | 8th Week
  Changes from baseline The Oswestry Disability Index (ODI) is a validated, 10-point patient-reported outcome questionnaire. The final score/index ranges from 0-100. A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound.

SECONDARY OUTCOMES:
Body Shape Questionnaire | 8th Week
  Changes from baseline the Body shape questionnaire is a self-reported measurement of body shape concerns designed for women to measure concerns about body image problems. The questionnaire has 34 items scored from 1 to 6 points. The overall total score range is between 34 to 204.
Double Leg lowering test | 8th Week
  Changes from baseline Double leg lowering test is used to assess abdominal muscles and the ability of muscles to maintain the posterior pelvic tilting position against the load. In this test Both legs are raised to a 90-degree angle (vertically) while keeping the upper body flat on the floor. The score is the angle of the legs in degrees from the floor. Total score ranges from 0 to 90 degrees, where 0 degree corresponds to excellent and 90 degrees is for very poor.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Ehsan, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Attock Hospital (Private) Limited, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No